CLINICAL TRIAL: NCT02491541
Title: A Single-centre, Randomized, Double-blind, Parallel Control, Phase 3 Study to Evaluate the Safety and Immunogenicity of a Rabies Vaccine (Vero Cell) for Human Use in Healthy Chinese Subjects Aged 10-60 Years
Brief Title: A Phase 3 Clinical Trial for a Rabies Vaccine (Vero Cell) for Human Use in Healthy Chinese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20120002
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Changchun Werersai (Experimental): A rabies vaccine (Vero Cell) for human use produced by Changchun Werersai Biotech Pharmaceutical Co., Ltd.
  Interventions: Biological: Changchun Werersai
- Jilin Maifeng (Active Comparator): A rabies vaccine (Vero Cell) for human use produced by Jilin Maifeng Biotech Pharmaceutical Co., Ltd.
  Interventions: Biological: Jilin Maifeng

INTERVENTIONS:
Biological: Changchun Werersai — A rabies vaccine (Vero Cell) for human use produced by Changchun Werersai Biotech Pharmaceutical Co., Ltd.
  1.0 ml experimental vaccine on day 0,3,7,14,28
  Arms: Changchun Werersai
Biological: Jilin Maifeng — A rabies vaccine (Vero Cell) for human use produced by Jilin Maifeng Biotech Pharmaceutical Co., Ltd.
  1.0 ml comparator vaccine on day 0,3,7,14,28
  Arms: Jilin Maifeng

SUMMARY:
The purpose of this single-centre, randomized, double-blind, parallel control, phase 3 study is to evaluate the safety and immunogenicity of a rabies vaccine (Vero Cell) for human use in healthy Chinese subjects aged 10-60 years, according to the Essen methods (1-1-1-1-1) vaccination.

DETAILED DESCRIPTION:
There will be two immunization arms. 1200 healthy subjects will be randomly assigned (1:1) to receive an experimental vaccine or a parallel comparator vaccine. All of them will be received five doses of rabies vaccine at day 0,3,7,14,28 according to the traditional Essen methods (1-1-1-1-1) vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 10 to 60 years old
* Subjects or legal guardians can and will comply with the requirements of the protocol
* Subjects or legal guardians are able to understand and sign the informed consent
* Healthy subjects judged from medical history after investigator's inquiry
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Female in lactation or pregnancy, or plan to be pregnant during the study period
* Subject who has allergic history to any vaccine or other medicines
* Subject who has injury history by dogs or other mammals and has been vaccinated with rabies vaccine
* Subject who has serious adverse reaction history after vaccination such as allergies, hives, difficulty in breathing, angioedema or abdominal pain
* Subject with congenital malformation, developmental disorder or serious chronic disease
* Subject with autoimmune diseases or immunodeficiency
* Subject with asthma, unstable over the past two years requiring emergency treatment, hospitalization, intubation, oral or intravenous corticosteroids
* Subject with diabetes (Type I or II) excluding gestational diabetes
* Subject with thyroidectomy history, or require treatment in the past 12 months due to thyroid disease
* Subject with severe angioedema in the past 3 years or require treatment in the past 2 years
* Subject with hypertension and with a blood pressure exceeding 145/95 mmHg at enrollment time
* Subject with coagulation abnormalities diagnosed by doctors (such as clotting factor deficiency, coagulation disorders, platelet disorder) or obvious bruises or blood clotting disorder
* Subject with cancer, or has been treated in active cancer period or not clearly cured, or may recur during the study period
* Subject with epilepsy, excluding those alcohol epilepsy within three years before quitting drinking or those do not need treatment in the past 3 years
* Asplenia, functional asplenia, without a spleen or removal of the spleen caused by any situation
* Guillain-Barre syndrome
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of other research medicine/vaccine in last 30 days
* Any prior administration of any attenuated live vaccine in last 30 days
* Any prior administration of subunit or inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Ongoing anti-tuberculosis prevention or treatment
* Subject who cannot comply with the trial requirements, or with mental illness/ dual-stage affective psychosis in the past or at present; or has not been controlled and needs to take psychiatric drugs the past 2 years; or with suicidal tendencies in the past 5 years
* Any medical, psychological, social or other condition judged by investigator, that may interfere subject's compliance with the protocol or signature on informed consent

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Positive seroconversion rate of serum rabies virus neutralizing antibody 42 days after full vaccination | 42 days after full vaccination

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) of serum rabies virus neutralizing antibody 42 days after full vaccination | 42 days after full vaccination
Positive seroconversion rate of serum rabies virus neutralizing antibody 14 days after full vaccination | 14 days after full vaccination
Geometric mean concentration (GMC) of serum rabies virus neutralizing antibody 14 days after full vaccination | 14 days after full vaccination
Incidence of local and systemic adverse reactions during safety observation period after each vaccination | 0-7 days after each vaccination and 8-28 days after the fifth vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Xinyi Center for Disease Control and Prevention, Xuzhou, Jiangsu, China